CLINICAL TRIAL: NCT06154941
Title: Clinical Evaluation of Giomer Based Varnish Versus CPP-ACP Varnish in the Management of Dentin Hypersensitivity: a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yomna sayed khallaf, lecturer at faculty of dentistry Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Giomer-CPPACP-Varnish
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giomer based Varnish (Experimental)
  Interventions: Procedure: Giomer Varnish
- CPP-ACP based varnish (Active Comparator)
  Interventions: Procedure: CPP-ACP varnish

INTERVENTIONS:
Procedure: Giomer Varnish — A light-cured Giomer varnish for prolonged hypersensitivity relief. Seals and protects exposed dentinal tubules to prevent pain. Ideal for patients experiencing loss of enamel, gingival recession
  Arms: Giomer based Varnish
Procedure: CPP-ACP varnish — CPP binds to oral surfaces such as teeth, dentin, oral mucosa and biofilm. CPP-ACP Varnish delivers bioavailable calcium and phosphate ions to occlude dentinal tubules treating dentin hypersensitivity
  Arms: CPP-ACP based varnish

SUMMARY:
Dentin hypersensitivity is a drastic problem, which threaten many dental patients. According to the last published systematic review and meta analysis at 2019, the prevalence of dentin hypersensitivity is being 33.5% among the population. Moreover, it was determined that young adults with age range from 18 to 44 years exhibited high percentage (43.9%) of such problem

DETAILED DESCRIPTION:
Several approaches to dentin hypersensitivity treatment were proposed to interfere, whether transiently or permanently, with the hydrodynamic theory. These approaches include root coverage and the use of lasers, ions, dentinal sealants, and occluding and nerve depolarization agents, chosen according to the primary cause. There are two major strategies in managing DH; the first is nerve desensitization, and the second is the physical occlusion of the patent tubule. The second approach can be carried out through a wide range of treatment modalities, including the use of proteins, salts or ions to plug the tubules. Many agents introduced are capable of sealing dentinal tubules, and can be used to reduce sensitivity. Of these agents are CPP-ACP varnish and the newly introduced giomer based varnish wilth S-PRG technology

ELIGIBILITY:
Inclusion Criteria:

* Participants of both genders aged 18 to 40 years with good oral hygiene, suffering from pain due to dentin hypersensitivity in at least one tooth

Exclusion Criteria:

* Taking desensitizing treatment in the last 6 months. (It affects the outcome)

  * Taking anti-inflammatory drugs. (It affects the hypersensitivity perception)
  * Pregnant females. ( They complain from nausea and repeated vomiting attacks)
  * Smokers. (Smoking will affect the oral hygiene and periodontal health)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
evaporative test | Immediately postoperative, after 1,3 and 6 months
  using an air blast from a conventional dental unit air-water syringe for 5 seconds.
Thermal Test | Immediately postoperative, after 1,3 and 6 months
  using anaesthetic carpule kept in the refrigerator at 4oC for at least 24 hours till it became ice then it is removed from refrigerator immediately before testing .
Tactile test | Immediately postoperative, after 1,3 and 6 months
  using the tip of a sharp explorer (number 3) to gently scratch the exposed cervical surface in an apico-coronal direction with short strokes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt